CLINICAL TRIAL: NCT05056259
Title: Usefulness of 18F-FDG PET/CT in the Initial Staging and Surveillance of Endometrial Cancer Patients
Acronym: PET/CT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya Abdel-Baset Ahmed Ali Alsanory, Resident in nuclear medicine departement (South Egypt Cancer institute), Assiut University
Other Study IDs: 18F-FDG PET/CT
Record Dates: First submitted 2021-09-15; First posted 2021-09-24 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- newly diagnosed endometrial cancer
  Interventions: Device: 18F-FDG PET/CT
- Recurrent cases of endometrial cancer
  Interventions: Device: 18F-FDG PET/CT

INTERVENTIONS:
Device: 18F-FDG PET/CT — The PET/CT procedure will be performed according to the institutional standard with 18F-FDG (0.8-1.2 mCi /kg) injection following 6 h fasting. Blood glucose was controlled to be <150 mg/dl. PET/CT from the vertex to the middle femur will be obtained 60 min after FDG injection.
  MDCT examination without IV contrast will be done for attenuation correction and anatomic localization followed by PET images from the skull vault to the mid-thigh region.
  Images of CT and corresponding functional PET images are displayed in axial, coronal and sagittal planes.
  PET/CT data will include tumor size and extension, LN invasion& distant metastasis SUVmax will be calculated for all positive lesions, Metabolic parameters including SUVmax, SUVmean, TLG & MTV will be calculated for primary tumor.
  Data of PET will be compared with other diagnostic imaging and postoperative pathologic data.

SUMMARY:
1. To assess the value of 18F-FDG PET/CT in the initial staging and detection of recurrent cases of endometrial cancer.
2. To determine correlation between PET/CT derived parameters including SUVmax, TLG and MTV and clinic-pathological patient characteristics.
3. To detect local and distant recurrence after therapy.

DETAILED DESCRIPTION:
Endometrial cancer (EC) is one of the most common gynaecological malignancies worldwide.The incidence rate of uterine cancer in Egypt was 4.1 per 100,000.

The standard surgery consists of laparotomy, hysterectomy, and bilateral salpingo-oophorectomy. Maximal surgical cytoreduction is recommended for advanced EC. Prognostic impact of complete lymphadenectomy remains controversial, especially in early- stage disease.

With the aim of predicting extrauterine disease pre-operatively and optimizing surgical planning, several techniques have been evaluated, including 18F-fluoro-2-deoxyglucose (18F-FDG) positron emission tomography/computed tomography (PET/CT). PET /CT can be used to effectively and accurately diagnose EC pelvic lymph node metastasis and distant metastasis. It has great value in clinical staging, judging prognosis, diagnosing recurrence.

Radiomics analysis of the uterine primary tumor on pre-operative 18F-FDG PET images may help predict the presence of metastatic nodes, thus reducing false-negative results and increasing the sensitivity of the technique. The maximum standard uptake value (SUVmax), metabolic tumor volume (MTV) and total glycolysis (TLG) of primary lesions are significantly correlated with pathological tissue grading. Previous studies on metabolic parameters of primary lesions examined by 18F-FDG PET/CT for endometrial cancer mainly focused on SUVmax, However, SUVmax can only reflect the functional metabolic degree of the point. It cannot assess the overall metabolic situation of tumor. MTV and TLG can more comprehensively measure the glucose metabolic activity of tumor cells with more clinical value in reflecting the malignancy degree of tumor.

ELIGIBILITY:
Inclusion Criteria:

* Patients proved to have endometrial cancer by curettage or hysteroscopy.
* Patients accepted surgery treatment, without anti-tumor and hormone therapy before surgery.
* Ability to stay still for the duration of the PET/CT scan (~15 minutes).
* Ability of the patient (or his/her guardian) to sign informed consent.

Exclusion Criteria:

* Patients who recieved neoadjuvant therapy before PET/CT.
* Patients with tumors other than endometrial cancer.
* Pregnancy.
* Inability to give informed consent.
* Inability to stay still for the duration of the scan.
* Claustrophobia

Min Age: 30 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Any patient proved to have endometrial cancer by curettage or hysteroscopy.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
To evaluate the correlation between metabolic parameters of primary lesions of endometrial cancer examined by 18F-FDG PET/CT and clinic-pathological features. | baseline
  Analysis of metabolic parameters and correlation between it and histopathology

SECONDARY OUTCOMES:
To evaluate diagnostic accuracy of PET/CT in the identification of EC stages | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Hanan Gamaleldin Mostafa, M.D, Study Chair — Professor; Esraa Roshdey Hassan, M.D, Study Director — Doctor

REFERENCES:
- [Background] Ferlay J, Soerjomataram I, Dikshit R, Eser S, Mathers C, Rebelo M, Parkin DM, Forman D, Bray F. Cancer incidence and mortality worldwide: sources, methods and major patterns in GLOBOCAN 2012. Int J Cancer. 2015 Mar 1;136(5):E359-86. doi: 10.1002/ijc.29210. Epub 2014 Oct 9. PMID 25220842
- [Background] Miller KD, Nogueira L, Mariotto AB, Rowland JH, Yabroff KR, Alfano CM, Jemal A, Kramer JL, Siegel RL. Cancer treatment and survivorship statistics, 2019. CA Cancer J Clin. 2019 Sep;69(5):363-385. doi: 10.3322/caac.21565. Epub 2019 Jun 11. PMID 31184787
- [Background] Alshahrani S, Soliman AS, Hablas A, Ramadan M, Meza JL, Remmenga S, Seifeldein IA, Chamberlain RM. Changes in Uterine Cancer Incidence Rates in Egypt. Obstet Gynecol Int. 2018 Jun 14;2018:3632067. doi: 10.1155/2018/3632067. eCollection 2018. PMID 30013598
- [Background] Gadducci A, Cosio S, Landoni F, Maggino T, Zola P, Sostegni B, Bellicini A, Fuso L, Cristofani R, Sartori E. Adjuvant treatment and analysis of failures in patients with high-risk FIGO Stage Ib-II endometrial cancer: an Italian multicenter retrospective study (CTF study). Gynecol Oncol. 2014 Jul;134(1):29-35. doi: 10.1016/j.ygyno.2014.04.008. Epub 2014 Apr 24. PMID 24769176
- [Background] Benedetti Panici P, Basile S, Salerno MG, Di Donato V, Marchetti C, Perniola G, Palagiano A, Perutelli A, Maneschi F, Lissoni AA, Signorelli M, Scambia G, Tateo S, Mangili G, Katsaros D, Campagnutta E, Donadello N, Greggi S, Melpignano M, Raspagliesi F, Cormio G, Grassi R, Franchi M, Giannarelli D, Fossati R, Torri V, Croce C, Mangioni C. Secondary analyses from a randomized clinical trial: age as the key prognostic factor in endometrial carcinoma. Am J Obstet Gynecol. 2014 Apr;210(4):363.e1-363.e10. doi: 10.1016/j.ajog.2013.12.025. Epub 2013 Dec 19. PMID 24361787
- [Background] Crivellaro C, Landoni C, Elisei F, Buda A, Bonacina M, Grassi T, Monaco L, Giuliani D, Gotuzzo I, Magni S, Di Martino G, Delle Marchette M, Guerra L, Landoni F, Fruscio R, Messa C, De Bernardi E. Combining positron emission tomography/computed tomography, radiomics, and sentinel lymph node mapping for nodal staging of endometrial cancer patients. Int J Gynecol Cancer. 2020 Mar;30(3):378-382. doi: 10.1136/ijgc-2019-000945. Epub 2020 Feb 19. PMID 32079712
- [Background] Gai QZ, Lv YB, Li GY, Zhang DQ, Gao Z, Fang XH. Value of metabolic parameters of primary lesions examined by 18F-FDG PET/CT for endometrial cancer in preoperative evaluation. Eur Rev Med Pharmacol Sci. 2021 Mar;25(6):2493-2502. doi: 10.26355/eurrev_202103_25412. PMID 33829435
- [Background] De Bernardi E, Buda A, Guerra L, Vicini D, Elisei F, Landoni C, Fruscio R, Messa C, Crivellaro C. Radiomics of the primary tumour as a tool to improve 18F-FDG-PET sensitivity in detecting nodal metastases in endometrial cancer. EJNMMI Res. 2018 Aug 22;8(1):86. doi: 10.1186/s13550-018-0441-1. PMID 30136163
- [Background] Rao L, Wang X, Zong Z, Chen Z, Shi X, Yi C, Zhang X, Yang Z. PET-CT for Evaluation of Spleen and Liver 18F-FDG Diffuse Uptake Without Lymph Node Enlargement in Lymphoma. Medicine (Baltimore). 2016 May;95(20):e3750. doi: 10.1097/MD.0000000000003750. PMID 27196500
- [Background] Husby JA, Reitan BC, Biermann M, Trovik J, Bjorge L, Magnussen IJ, Salvesen OO, Salvesen HB, Haldorsen IS. Metabolic Tumor Volume on 18F-FDG PET/CT Improves Preoperative Identification of High-Risk Endometrial Carcinoma Patients. J Nucl Med. 2015 Aug;56(8):1191-8. doi: 10.2967/jnumed.115.159913. Epub 2015 Jun 4. PMID 26045311